CLINICAL TRIAL: NCT03552484
Title: CarePSP: Care Where It Counts - Interdisciplinary Home Visits for PSP-Related Disorders
Brief Title: In-Home Care for Patients With PSP and Related Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 17101005; 633-2016-10 (Other Grant/Funding Number: CurePSP)
Record Dates: First submitted 2018-04-16; First posted 2018-06-11 (Actual); Results first posted 2024-04-01 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-10

CONDITIONS: Progressive Supranuclear Palsy; Dementia With Lewy Bodies; Multiple System Atrophy; Corticobasal Syndrome; Atypical Parkinson Disease
MeSH Terms: conditions — Supranuclear Palsy, Progressive; Lewy Body Disease; Multiple System Atrophy; Corticobasal Degeneration; Parkinson Disease, Familial, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home Visit Arm (Active Comparator): Participants and their caregivers, when available, will be asked to participate in four study visits, which will involve in-home clinical assessments, a needs assessment, and completion of some questionnaires. Additional information will be obtained from patients' routine medical records: their medical and medication history, family history, neurological examination findings, and office visit records.
  [Completion of Home Visit Program]
  Interventions: Behavioral: Home Visit Program
- Usual Care Arm (Active Comparator): Participants and their caregivers, when available, will be asked to complete an initial online survey. Twelve months later, patients (and caregivers, if available) will be asked to complete an online follow-up survey.
  [Completion of Usual Care/Online Survey]
  Interventions: Behavioral: Usual Care/Online Survey

INTERVENTIONS:
Behavioral: Home Visit Program — Informed consent discussion, documentation; UPDRS I-IV, medical history, vitals, medication reconciliation, patient medical history and comorbidities; home safety assessment; psychosocial assessment of dyad, resource utilization questionnaire, caregiver medical history and comorbidities, MCSI; patient and caregiver short MoCA, satisfaction surveys, EQ5D; counseling, summarizing plan of care
  Arms: Home Visit Arm
Behavioral: Usual Care/Online Survey — Patients and caregivers, if available, will be asked to complete an online survey that asks about demographics, disease history, resource utilization, and unmet needs. The will be asked to complete a follow-up survey 12 months after completion of the initial survey.
  Arms: Usual Care Arm

SUMMARY:
Progressive Supranuclear Palsy and related disorders (PRD) are debilitating, costly, and understudied conditions. Improving access to comprehensive, specialized, in-home patient care offers the potential to minimize the downward spiral of morbidity and preventable healthcare utilization. The aim of this study is to test whether and to what degree an interdisciplinary home visit program will improve patient- and caregiver-reported outcomes, and to identify unmet needs in this population.

DETAILED DESCRIPTION:
Participants can elect to complete either the Home Visit Arm of the study or the Usual Care Arm of the study.

Home Visit Arm:

This interdisciplinary home visit program consists of 4 visits to patients' homes over the course of one year from a team of a movement disorders doctor, a nurse, a research coordinator, and a social worker. The team will come to a patient's home and assess the needs of both the patient and caregiver (if present), and connect the patient with any needed services. These visits can replace or be in addition to seeing another movement disorders doctor.

Usual Care Arm:

The information collected from the home visit participants will be compared to data collected from participants who elect to complete the usual care arm of the study. These participants and their caregivers (if available) will be invited to complete an online version of the survey. They will be contacted 12 months after their initial completion of the survey to complete a follow-up survey.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be those diagnosed with progressive supranuclear palsy, multiple system atrophy, corticobasal syndrome , Dementia with Lewy Bodies (DLB), or atypical parkinsonism without mention of idiopathic Parkinson's disease.
* Subjects must be English speaking.

Additional Inclusion Criteria For the Home Care Arm:

* Each subject must either 1) be willing and able to provide written, informed consent for the study, and for whom capacity to consent will be assessed, or 2) if unable to provide informed consent due to lack of capacity, a caregiver is able to provide informed consent and the subject provides assent to participation.
* Subjects must be homebound according to the Medicare definition: "Leaving your home isn't recommended because of your condition; your condition keeps you from leaving home without help (such as using a wheelchair or walker, needing special transportation, or getting help from another person); leaving home takes a considerable and taxing effort." (http://www.medicare.gov/pubs/pdf/10969.pdf)
* Subjects reside in Chicago at the time of Visit 1.
* The Subject must reside independently at the time of Visit 1.
* Subjects have one or more of the following criteria: fluctuation, multi-morbidity, mismanages medication, cognitive impairment, symptoms of depression and/or anxiety, high risk for re-hospitalization, high risk for nursing facility admission, suspected elder abuse, recent history of increased falls in home, caregiver burnout suspected
* Ability to participate in the research study as deemed by the Principal Investigator.

Additional Inclusion Criteria For the Usual Care Arm:

* Independent access to an internet-connected computer in order to complete online survey
* Valid email address
* Each subject must review and acknowledge their ability to provide informed consent for the study via the first screen of the online survey

Exclusion Criteria:

* Diagnosis of idiopathic Parkinson's Disease
* Diagnosis of another neurodegenerative disease
* Subjects with active psychosis or exhibiting symptoms of a severe psychiatric disorder

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jori Fleisher, MD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Home Visit Arm: Participants will be asked to participate in four study visits, which will involve in-home clinical assessments, a needs assessment, and completion of some questionnaires. Additional information will be obtained from patients' routine medical records: their medical and medication history, family history, neurological examination findings, and office visit records.
  [Completion of Home Visit Program]
  Home Visit Program: Informed consent discussion, documentation; UPDRS I-IV, medical history, vitals, medication reconciliation, patient medical history and comorbidities; home safety assessment; psychosocial assessment of dyad, resource utilization questionnaire, caregiver medical history and comorbidities, MCSI; patient and caregiver short MoCA, satisfaction surveys, EQ5D; counseling, summarizing plan of care
  In the event that a patient is unable to answer the survey questions on their own but has a knowledgeable caregiver who can answer on their behalf, the caregiver can complete the survey as the patient's proxy, answering questions AS the patient.
  All counts include PATIENTS only
- Usual Care Arm (NOT RANDOMIZED): Patients will be asked to complete an initial online survey. Twelve months later, patients will be asked to complete an online follow-up survey.
  [Completion of Usual Care/Online Survey]
  Usual Care/Online Survey: Patients will be asked to complete an online survey that asks about demographics, disease history, resource utilization, and unmet needs. The will be asked to complete a follow-up survey 12 months after completion of the initial survey.
  In the event that a patient is unable to answer the survey questions on their own but has a knowledgeable caregiver who can answer on their behalf, the caregiver can complete the survey as the patient's proxy, answering questions AS the patient.
  All counts include PATIENTS only
Period: Overall Study
Arm/Group | Home Visit Arm | Usual Care Arm (NOT RANDOMIZED)
Started | 20 | 36
Completed | 14 | 16
Not Completed | 6 | 20
Not completed — Death | 6 | 4
Not completed — Lost to Follow-up | 0 | 16

BASELINE CHARACTERISTICS:
Population: Two participants in the usual care arm signed the informed consent but did not complete any surveys, including demographic information, explaining the difference between the 36 in the protocol and participant flow modules, and 34 here.
Groups:
- Home Visit Arm: Participants will be asked to participate in four study visits, which will involve in-home clinical assessments, a needs assessment, and completion of some questionnaires. Additional information will be obtained from patients' routine medical records: their medical and medication history, family history, neurological examination findings, and office visit records.
  [Completion of Home Visit Program]
  Home Visit Program: Informed consent discussion, documentation; UPDRS I-IV, medical history, vitals, medication reconciliation, patient medical history and comorbidities; home safety assessment; psychosocial assessment of dyad, resource utilization questionnaire, caregiver medical history and comorbidities, MCSI; patient and caregiver short MoCA, satisfaction surveys, EQ5D; counseling, summarizing plan of care
- Usual Care Arm (NOT RANDOMIZED): Participants will be asked to complete an initial online survey. Twelve months later, patients will be asked to complete an online follow-up survey.
  [Completion of Usual Care/Online Survey]
  Usual Care/Online Survey: Patients will be asked to complete an online survey that asks about demographics, disease history, resource utilization, and unmet needs. The will be asked to complete a follow-up survey 12 months after completion of the initial survey.
- Total: Total of all reporting groups
Arm/Group | Home Visit Arm | Usual Care Arm (NOT RANDOMIZED) | Total
Number analyzed (Participants) | 20 | 34 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 17 | 28 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.2 (8.1) | 71.7 (7.7) | 72.3 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 28
  Male | 7 | 19 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 20 | 30 | 50
  Unknown or Not Reported | 0 | 3 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 17 | 33 | 50
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 34 | 54
Diagnosis [Count of Participants; unit: Participants]
  Progressive Supranuclear Palsy | 8 | 23 | 31
  Multiple System Atrophy | 7 | 5 | 12
  Corticobasal Syndrome | 3 | 2 | 5
  Atypical parkinsonism | 2 | 4 | 6
Self-reported homebound status [Count of Participants; unit: Participants] — Meets Centers for Medicare and Medicaid services definition of homebound, namely, 1) requires a considerable and taxing effort to leave the home due to medical condition, and 2) requires EITHER an assistive device, assistive transportation, or a care partner or other accompanying individual to assist with leaving the home
  Participants | 20 | 29 | 49

OUTCOME MEASURES:

1. Primary Outcome: Change in Patient Quality of Life as Measured by the EuroQol 5-D (EQ-5D) Scale Between Baseline (Visit 1) and 1 Year (Visit 4)
Description: This scale is a brief, 6-item instrument measuring five specific domains of health-related quality of life (mobility, self-care, activities of daily living, anxiety/depression, pain/discomfort) and overall well-being. Items are scored on a 1-5 scale, with 5 indicating the highest level of perceived problems. Scores at Visits 1 and 4 will be compared.
Time Frame: 1 year
Population: In the home visit arm, six patients died between visits 1 and 4, yielding a cohort of 14 patients available to complete surveys at visit 4.
  In the usual care arm, only sixteen participants responded to at least one survey at month 12; the remainder were lost to follow-up despite multiple attempts to reach them via email over a period of weeks.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Home Visit Arm | Usual Care Arm (NOT RANDOMIZED)
Number analyzed (Participants) | 14 | 16
units on a scale
  Mobility | 1 [0 to 2] | 0.5 [0 to 1]
  Self-care | 0.5 [0 to 2] | 0 [-1 to 3]
  Activities of daily living | 1 [0 to 3] | 0 [-1 to 2]
  Anxiety/depression | 0 [-1 to 2] | 0 [-1 to 2]
  Pain/discomfort | 0 [-3 to 4] | 0 [-2 to 1]
Statistical Analysis 1: Comparison: Home Visit Arm vs Usual Care Arm (NOT RANDOMIZED); Within-group paired t-tests and between-group paired t-tests; Test type: Superiority; p = 0.59, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.05

2. Primary Outcome: Change in Overall Quality of Life as Measured by the EuroQol 5-D (EQ-5D) Scale Visual Analog Scale Item Between Baseline (Visit 1) and 1 Year (Visit 4)
Description: This item is a 0-100 point visual analog scale for rating overall quality of life where 0 is "the worst" and 100 "the best health you can imagine". Scores at Visits 1 and 4 will be compared.
Time Frame: 1 year
Population: In the home visit arm, six patients died between visits 1 and 4, yielding a cohort of 14 patients available to complete surveys at visit 4. Five of the 14 did not complete the visual analog scale.
  In the usual care arm, only sixteen participants responded to at least one survey at month 12, however six of the 16 did not complete the visual analog scale; the remainder were lost to follow-up despite multiple attempts to reach them via email over a period of weeks.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Home Visit Arm | Usual Care Arm (NOT RANDOMIZED)
Number analyzed (Participants) | 9 | 10
score on a scale | -1.43 (38.85) | 4.81 (23.82)
Statistical Analysis 1: Comparison: Home Visit Arm vs Usual Care Arm (NOT RANDOMIZED); Test type: Superiority; p = 0.59, t-test, 2 sided — Between-group comparison; Mean Difference (Final Values) = -1.43

3. Secondary Outcome: Change in Caregiver Strain as Measured by the Multidimensional Caregiver Strain Index (MCSI) Between Baseline (Visit 1) and 1 Year (Visit 4)
Description: An 18-item tool measuring subjective response to stressors. Respondents are asked about the frequency with which items apply, ranging from "never" to "all of the time" on a 5 point scale. The range is from 0 to 72, where higher scores indicate higher levels of caregiver strain, and scores in the 20-29 range are categorized as "moderate" strain, and scores 30 or higher are categorized as severe strain. Scores at Visits 1-4 will be compared.
Time Frame: 1 year
Population: Nine home visit caregivers completed surveys at baseline AND visit 4/twelve months; ten usual care caregivers completed surveys at baseline and twelve months. The remainder of participants did not have caregivers available at the time of home visit or survey completion, respectively.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Home Visit Arm: Caregivers of home visit participants, when available, will be asked to participate in four study visits.
- Usual Care Arm (NOT RANDOMIZED): Caregivers of usual care participants, if available, completing an online survey at baseline and twelve months later.
Arm/Group | Home Visit Arm | Usual Care Arm (NOT RANDOMIZED)
Number analyzed (Participants) | 9 | 10
score on a scale | 0.44 (5.77) | 2.3 (9.46)
Statistical Analysis 1: Comparison: Home Visit Arm vs Usual Care Arm (NOT RANDOMIZED); Test type: Superiority; p = 0.62, t-test, 2 sided — Between-group comparison of change in Multidimensional Caregiver Strain Index; Mean Difference (Final Values) = 0.44

4. Other Pre Specified Outcome: Patient Satisfaction With the Home Visit Program as Measured by the Client Satisfaction Inventory- Short Form (CSI-SF)
Description: A 9-item instrument developed within the field of social work to assess client satisfaction with multidisciplinary programs like the home visit program in this study. Each item is scored on a 1-7 scale, for a total possible raw score of 7-63, scaled to 0-100% of the possible score, with higher scores indicating greater client satisfaction. This measure will be completed at our last home visit (Visit 4).
Time Frame: 1 year
Population: 14 patients completed visit 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Home Visit Participants - Patients: Homebound individuals with a diagnosis of progressive supranuclear palsy, multiple system atrophy, corticobasal syndrome, or atypical parkinsonism who consented to four home visits over one year; participants completed the nine-item Client Satisfaction Inventory-Short Form about the multidisciplinary care they received in the home visit intervention at the time of home visit 4
Arm/Group | Home Visit Participants - Patients
Number analyzed (Participants) | 14
score on a scale | 100 [77.8 to 100]

5. Other Pre Specified Outcome: Caregiver Satisfaction With the Home Visit Program as Measured by the Client Satisfaction Inventory- Short Form (CSI-SF)
Description: as for outcome 4
Time Frame: 1 year
Population: 10 caregivers completed the surveys at visit 4
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Home Visit Participants - Caregivers: Homebound individuals with a diagnosis of progressive supranuclear palsy, multiple system atrophy, corticobasal syndrome, or atypical parkinsonism who consented to four home visits over one year; caregivers of homebound individuals completed the nine-item Client Satisfaction Inventory-Short Form about the multidisciplinary care they received in the home visit intervention at the time of home visit 4
Arm/Group | Home Visit Participants - Caregivers
Number analyzed (Participants) | 10
score on a scale | 98 [87.0 to 100]

ADVERSE EVENTS:
Time Frame: 1 year
Description: Survey data
Arm/Group | Home Visit Arm | Usual Care Arm (NOT RANDOMIZED)
All-Cause Mortality (participants affected / at risk) | 6/20 | 4/36
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/36
Other Adverse Events (participants affected / at risk) | 0/20 | 0/36

LIMITATIONS AND CAVEATS:
This was not a randomized trial and the "usual care"/control group was poorly defined and suffered from significant loss to follow-up. The usual care group was recruited via online survey and completed a battery of online surveys at baseline. One year later, the usual care participants received up to five emails at the email address initially provided upon enrollment. There was significant loss to follow-up with lack of response to emailed reminders.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03552484/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-18): https://cdn.clinicaltrials.gov/large-docs/84/NCT03552484/SAP_001.pdf